CLINICAL TRIAL: NCT00186810
Title: Allogeneic Stem Cell Transplantation From HLA/MLC Genotype Identical Donors for Patients With High Risk Sickle Cell Disease
Brief Title: Stem Cell Transplantation With Identical Donors for Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Gregory Hale, MD / Principal Investigator, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCALLO
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Sickle Cell Disease
Keywords: Anemia; Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia | interventions — Busulfan; Cyclophosphamide; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Busulfan, Cyclophosphamide, Horse ATG; Procedure: Allogeneic stem cell transplant

INTERVENTIONS:
Drug: Busulfan, Cyclophosphamide, Horse ATG — Transplant recipients received a myeloablative conditioning regimen of cyclophosphamide, Anti-Thymocyte Globulin (horse), and Busulfan. Cyclosporine and methotrexate were administered for GVHD prophylaxis.
Procedure: Allogeneic stem cell transplant — Allogeneic stem cell transplant Matched sibling donor transplant Cord blood transplant

SUMMARY:
This protocol studied the effect of administration of a myeloablative pretransplant preparative regimen followed by an infusion of donor stem cells in children with severe sickle cell disease. The donor graft consisted of bone marrow or cord blood derived from a genetically matched sibling.

The primary aim of the study was to evaluate how well the donated cells migrated to the bone marrow and begin producing healthy red blood cells, white blood cells and platelets (engrafted), how well the recipients immune system recovered, and assess any regimen related toxicities including a potentially life-threatening transplant related complication called graft-versus-host-disease or GVHD.

DETAILED DESCRIPTION:
The secondary objectives of this protocol evaluated the effect of this transplant procedure on the subsequent clinical course of patients with severe SCD. Specifically, to determine whether pre-transplant organ dysfunction (brain, heart, lung, kidney, liver, spleen, etc) resultant from sickle hemoglobinopathy can be reversed following this particular transplant procedure.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of severe' disease is denoted by one of the following:

* Previous central nervous system vaso-occlusive episode with or without residual neurologic findings or
* Frequent painful vaso-occlusive episodes with significant interference with normal life activities and which necessitates chronic transfusion therapy or
* Recurrent SCD chest syndrome events which necessitate chronic transfusion therapy.

Exclusion criteria:

* Patient with SCD chronic lung disease greater than or equal to stage 3
* Patient with severe renal dysfunction defined as creatinine clearance < 40 ml/min/1.73m2.
* Patient with severe cardiac dysfunction defined as echocardiogram shortening fraction < 25%.
* Patient with HIV infection.
* Pregnant or lactating.
* Patient with unspecified chronic toxicity that in the opinion of the Principal Investigator is serious enough to detrimentally affect the patient's capacity to tolerate SCT.
* Patient or patient's guardian(s) unable to understand the nature and risks inherent in the BMT process

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 1992-12; Primary Completion 2006-02 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To evaluate engraftment, GVHD, hematopoietic and immune reconstitution, and regimen-related mortality and morbidity in patients with severe sickle cell disease undergoing transplant using either HLA matched sibling bone marrow or cord blood grafts. | March 2007

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hale, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Dallas MH, Triplett B, Shook DR, Hartford C, Srinivasan A, Laver J, Ware R, Leung W. Long-term outcome and evaluation of organ function in pediatric patients undergoing haploidentical and matched related hematopoietic cell transplantation for sickle cell disease. Biol Blood Marrow Transplant. 2013 May;19(5):820-30. doi: 10.1016/j.bbmt.2013.02.010. Epub 2013 Feb 14. PMID 23416852
- See also: St. Jude Children's Research Hospital — http://www.stjude.org